CLINICAL TRIAL: NCT05491980
Title: Creating a Florida Cerebrovascular Disease Biorepository and Genomics Center
Brief Title: Florida Cerebrovascular Disease Biorepository and Genomics Center
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, James F. Meschia, Principal Investigator, Mayo Clinic
Other Study IDs: 22-002667
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Cerebrovascular Disease; Ischemic Stroke; Transient Ischemic Attack; Intracerebral Hemorrhage; Aneurysmal Subarachnoid Hemorrhage; Vascular Dementia; Anoxic Brain Injury; Unruptured Intracranial Aneurysm; Carotid Artery Stenosis Symptomatic; Asymptomatic Carotid Artery Stenosis; Non-Aneurysmal Perimesencephalic Subarachnoid Haemorrhage; Cerebral Venous Thrombosis; Moyamoya Disease; Fibromuscular Dysplasia; Subarachnoid Hemorrhage; Leukoaraiosis; Arteriovenous Fistula; Reversible Cerebral Vasoconstriction Syndrome; CADASIL
MeSH Terms: conditions — Cerebrovascular Disorders; Ischemic Stroke; Ischemic Attack, Transient; Cerebral Hemorrhage; Subarachnoid Hemorrhage; Dementia, Vascular; Hypoxia-Ischemia, Brain; Intracranial Thrombosis; Moyamoya Disease; Fibromuscular Dysplasia; Leukoaraiosis; Arteriovenous Fistula; CADASIL

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to create a state-wide biorepository and resource center for cerebrovascular diseases in Florida, which will include collecting medical history information and blood from subjects affected by cerebrovascular disease. The information and blood samples collected may be used in future research for the study of cerebrovascular disease and to learn about, prevent or treat other health problems.

ELIGIBILITY:
Inclusion Criteria:

• Affected subjects with diverse cerebrovascular conditions, including, but not limited to, ischemic stroke, transient ischemic attack (TIA), intracerebral hemorrhage (ICH), aneurysmal subarachnoid hemorrhage (aSAH), vascular dementia (VAD), anoxic brain injury, unruptured intracranial aneurysm (UIA), cavernous malformation, arteriovenous malformations (AVM), carotid and vertebral arterial dissections, symptomatic and asymptomatic cervical carotid artery atherosclerotic stenosis, non-aneurysmal perimesencephalic subarachnoid hemorrhage (naSAH), cerebral venous thrombosis (CVT), moyamoya disease, fibrosmuscular dysplasia (FMD), non-traumatic, angiography-negative subarachnoid hemorrhage, leukoaraiosis, arteriovenous fistula, reversible cerebral vasoconstriction syndrome (RCVS), and CADASIL.

Exclusion Criteria:

• All patients with the following known or suspected virulent microorganisms causing an active or latent infection will be excluded from the study:

* Human immunodeficiency virus (HIV);
* Any viral hepatitis;
* West Nile virus (WNV);
* Influenza virus;
* Tuberculosis (TB);
* Any bacteremia;
* Any fungemia;
* Any prionopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects identified with a history of cerebrovascular disease will be recruited from both the in-patient and outpatient services at Mayo Clinic Florida.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Stroke or TIA at 12 months | 1 year
  Number of participants to experience new diagnosis of TIA or stroke.

SECONDARY OUTCOMES:
Modified Rankin Scale | 1 year
  Measure of overall functional status

CONTACTS AND LOCATIONS:
Overall Officials: James Meschia, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials